CLINICAL TRIAL: NCT00860405
Title: Efficacy and Safety of 6 % Hydroxyethyl Starch 130/0.4 (Voluven®) vs. 5% HSA in Volume Replacement Therapy During Elective Open-heart Surgery in Paediatric Patients
Brief Title: Voluven® in Paediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HE06-001-C P4
Record Dates: First submitted 2009-02-27; First posted 2009-03-12 (Estimated); Results first posted 2011-09-19 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; Sodium Chloride; HES 130-0.4; Solutions; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Investigational drug: HES 130/0.4 (6%) in sodium chloride (Voluven®, solution for infusion)
  Interventions: Drug: HES 130/0.4 (6%) in sodium chloride (Voluven®, solution for infusion), Human serum albumin (HSA 50g/L)
- 2 (Active Comparator): Control drug: Human serum albumin (HSA 50g/L)
  Interventions: Drug: Human serum albumin (HSA 50g/L)

INTERVENTIONS:
Drug: HES 130/0.4 (6%) in sodium chloride (Voluven®, solution for infusion), Human serum albumin (HSA 50g/L) — Study medication will be given as part of the priming of the ECC and for plasma volume replacement after start of ECC up to the maximum dosage of 50 mL/kg body weight/day.
  Other Names: Voluven®
  Arms: 1
Drug: Human serum albumin (HSA 50g/L) — Human serum albumin (HSA 50g/L)
  Arms: 2

SUMMARY:
This study will compare the clinical efficacy and safety of Voluven® and Human Albumin during elective open-heart surgery in pediatric patients.

DETAILED DESCRIPTION:
In the past, human albumin has been widely accepted as the therapeutic "gold standard" in paediatric volume replacement therapy because of the physiological hypoproteinemia in newborns and infants. In adult patients, artificial colloids such as hydroxyethyl starch have replaced human albumin as first choice in many settings. This study will compare the clinical efficacy and safety of HES 130/0.4 (6%) in normal saline vs. HSA 50g/L in volume replacement therapy during elective open-heart surgery in paediatric patients. The hypothesis of this study is to demonstrate that HES 130/0.4 (6%) and HSA 50g/L are equivalent regarding efficacy and provide comparable safety during elective open-heart surgery in paediatric patients 2 to 12 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female paediatric patient, 2 to 12 years of age, suffering from congenital heart-disease and undergoing elective open-heart surgery requiring ECC;
* Signed parental written informed consent and patient assent where achievable

Exclusion Criteria:

* Known contraindication against scheduled concomitant medication;
* Total ECC volume < 400 mL;
* ASA > III

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Van der Linden, Professor, Principal Investigator — HUDERF - Hôpital Universitaire des Enfants Reine Fabiola; Hans Gombotz, Professor, Principal Investigator — AKh Allgemeines Krankenhaus der Stadt Linz GmbH
Locations (2):
- AKh Allgemeines Krankenhaus der Stadt Linz GmbH, Linz, Austria
- HUDERF - Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in paediatric care units of 2 hospitals in Austria and Belgium from March 2009 (FPI) until July 2010 and were followed up until August 2010 (LPO).
Pre-assignment Details: Participants were screened in paediatric care units of the participating 2 study sites in Austria and Belgium.
Groups:
- Voluven® Arm: 6% Hydroxyethylstarch 130/0.4, i.v. Voluven® rates were not to exceed 50 mL/kg/day; if additional study drug was required, 5% HSA was provided as rescue colloid.
- HSA 5% Arm (Comparison Group): Human Serum Albumin (HSA) 50g/L, i.v.
Period: Overall Study
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group)
Started | 31 | 30
Completed Treatment | 31 | 29
Day 28 Follow-up Performed | 31 | 29
Completed | 26 (completed overall study) | 26
Not Completed | 5 | 4
Not completed — Main reason: Follow-up data not complete | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group) | Total
Number analyzed (Participants) | 31 | 30 | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 5.2 (2.9) | 4.0 (2.0) | 4.6 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  Belgium | 20 | 20 | 40
  Austria | 11 | 10 | 21
Weight [Mean (Standard Deviation); unit: kg] | 18.2 (8.9) | 15.4 (4.4) | 16.9 (7.2)
Height [Mean (Standard Deviation); unit: cm] | 106.6 (16.8) | 101.3 (12.8) | 104.0 (15.1)

OUTCOME MEASURES:

1. Primary Outcome: Total Volume of Colloid Solution Required Intraoperatively
Description: Total volume of study drug plus rescue colloid, if applicable
Time Frame: Day 1 (intraoperatively)
Population: Per-protocol population (PP) = All patients in the Intention-to-treat (ITT) set without any major protocol violation.
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group)
Number analyzed (Participants) | 29 | 26
ml/kg | 36.6 (11.76) | 36.97 (11.86)
Statistical Analysis 1: Comparison: Voluven® Arm vs HSA 5% Arm (Comparison Group); The aim of the study was to prove equivalence, i.e. H0: μVoluven/μHSA ≤ 0.55 or μVoluven/μHSA ≥ 1.82 H1: 0.55 < μVoluven/μHSA < 1.82 where μVoluven was the mean infused volume of Voluven® and μHSA was the mean infused volume of HSA 5%; Test type: Non-Inferiority or Equivalence — Assuming a coefficient of variation of 0.363 and a desired power of 90 % with a type I level of 2.5 %, N=11 patients per treatment group were needed. The power was calculated by means of the software SAS, version 9.1.3, PROC POWER. Nevertheless, more patients were required for the assessment of safety, therefore 2 × 30 patients were planned to be included in this study; ANOVA — Null hypothesis tested by calculating a 2-sided 95% CI for ratio of LS-means μVoluven/μHSA based on ANOVA incl.treatment+centre as effects. If 95% CI was within equivalence range(0.55, 1.82), significant equivalence was concluded (Type I error: 2.5%); Primary endpoint specified + analysed for PP and ITT population. Confirmatory analysis based on PP population only, no adjustment for multiplicity; Ratio of LS-means = 0.98, 95% CI 2-sided [0.84 to 1.16] — Considered ratio: μVoluven/μHSA = LS-mean of Voluven®/LS-mean of HSA 5%

2. Secondary Outcome: Mean Arterial Pressure (MAP)
Description: Mean arterial pressure (MAP) from beginning of anaesthesia (baseline) until arrival on intensive care unit (ICU)
Time Frame: Beginning of anaesthesia (baseline) until arrival on intensive care unit (ICU)
Population: Per-protocol population (PP) = All patients in the ITT set without any major protocol violation
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group)
Number analyzed (Participants) | 29 | 26
mm Hg
  T0, Baseline | 64.1 (11.3) | 66.5 (12.5)
  T1, before ECC (Extracorporeal circulation) | 54.0 (7.4) | 51.3 (8.0)
  T2, after ECC | 56.6 (7.6) | 58.2 (9.7)
  T3, after skin closure | 61.2 (9.7) | 62.0 (9.9)
  T4, arrival on ICU | 65.3 (14.8) | 65.2 (8.8)

3. Secondary Outcome: Fluid Input
Description: Quantity of total fluids administered from beginning of anaesthesia until 2nd postop morning
Time Frame: 2 days
Population: Per-protocol population (PP) = All patients in the ITT set without any major protocol violation
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group)
Number analyzed (Participants) | 29 | 26
ml/kg | 246.8 (119.3) | 248.2 (105.8)

4. Secondary Outcome: Fluid Output
Description: Quantity of total fluids excreted or lost from beginning of anaesthesia until 2nd postop morning
Time Frame: 2 days
Population: Per-protocol population (PP) = All patients in the ITT set without any major protocol violation.
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group)
Number analyzed (Participants) | 29 | 26
ml/kg | 195.5 (95.7) | 181.1 (68.3)

5. Secondary Outcome: Fluid Balance
Description: Balance of total fluid input and total fluid output
Time Frame: 2 days
Population: Per-protocol population (PP) = All patients in the ITT set without any major protocol violation.
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group)
Number analyzed (Participants) | 29 | 26
ml/kg | 51.3 (47.5) | 67.1 (62.6)

6. Other Pre Specified Outcome: Calculated Perioperative Red Blood Cell (RBC) Loss
Description: Calculated perioperative RBC loss = Predicted blood volume1 × (hematocrit [baseline] - hematocrit [2nd postop morning]) + transfused RBC volume2;
  1. Predicted blood volume (mL) = 80 × body weight (kg)
  2. Transfused RBC volume = 0.7 × infused packed RBC
Time Frame: 2 days
Population: Safety Population (SAF) = All randomized patients treated with study drug.
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group)
Number analyzed (Participants) | 31 | 29
ml/kg | 14.4 (14.4) | 15.3 (15.5)

7. Other Pre Specified Outcome: Length of Stay on the Intensive Care Unit (ICU)
Description: Length of stay (number of days) on the intensive care unit (ICU).
Time Frame: From admission to ICU until discharge from ICU
Population: Safety Population (SAF) = All randomized patients treated with study drug.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group)
Number analyzed (Participants) | 31 | 29
Days | 3.1 [2.0 to 5.8] | 3.1 [2.3 to 6.9]

8. Other Pre Specified Outcome: Mortality
Description: Mortality was reported for the time period from screening until the end of follow-up.
Time Frame: From screening to end of follow-up
Population: Safety Population (SAF) = All randomized patients treated with study drug
Measure: Number; unit: Participants
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group)
Number analyzed (Participants) | 31 | 29
Participants | 0 | 0

9. Other Pre Specified Outcome: Acute Renal Failure (ARF)
Description: Acute renal failure was defined as a two fold increase in serum creatinine concentration over the value at baseline at any time after baseline.
Time Frame: From baseline until 2nd postop morning.
Population: Safety Population (SAF) = All randomized patients treated with study drug.
Measure: Number; unit: Participants
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group)
Number analyzed (Participants) | 31 | 29
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse event recording was performed throughout the study (from signing the informed consent until the follow-up visit at 28 days after discharge from operating room).
Description: Regular assessment by Pharmacovigilance and Safety Assessor
Arm/Group | Voluven® Arm | HSA 5% Arm (Comparison Group)
Serious Adverse Events (participants affected / at risk) | 11/31 | 7/29
Other Adverse Events (participants affected / at risk) | 30/31 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voluven® Arm (N=31) | HSA 5% Arm (Comparison Group) (N=29)
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1
Internal hernia (Gastrointestinal disorders) | 1 | 0
Device breakage (General disorders) | 1 | 0
Medical device complication (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 2
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Post procedural pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Circulatory collapse (Vascular disorders) | 0 | 1
Haemodynamic instability (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voluven® Arm (N=31) | HSA 5% Arm (Comparison Group) (N=29)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 1
Nodal rhythm (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 7 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 13 | 9
Device occlusion (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 3
Exposure to contaminated device (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Infusion site urticaria (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 2 | 1
Aspergillosis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Enterobiasis (Infections and infestations) | 0 | 1
H1n1 Influenza (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 4
Lobar pneumonia (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Post procedural pneumonia (Infections and infestations) | 2 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin candida (Infections and infestations) | 1 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Dilutional coagulopathy (Injury, poisoning and procedural complications) | 1 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 7 | 6
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 4
Blood lactic acid increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 1
Enterovirus test positive (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Venous oxygen saturation decreased (Investigations) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 17 | 13
Hyperlactacidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 10 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 8 | 8
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 1
Phrenic nerve paralysis (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 6 | 3
Anxiety (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 2 | 2
Haematuria (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Reproductive system and breast disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haemodynamic instability (Vascular disorders) | 4 | 4
Hypotension (Vascular disorders) | 10 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications are subject to a prior review of Fresenius Kabi and may only be made in a neutral and anonymous form within the respective circles of experts. Fresenius Kabi shall give its comments, if applicable, within 30 days after having received the respective manuscript. Manuscripts should be submitted for publication within 2 years following the final report.